CLINICAL TRIAL: NCT02994004
Title: Medical Decision-making Under Budgetary Constraint: an fMRI Study
Brief Title: Exploring Medical Decisions Using Functional MRI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8989
Record Dates: First submitted 2016-09-05; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2014-07

CONDITIONS: F-MRI Brain Imaging Data
Keywords: Hospital, medical decision-making, role conflict, f-MRI

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
Hospital physicians are increasingly facing budgetary constraints that might have an impact on individual medical decisions (i.e. diagnostic or therapeutic decisions). This might translate into role conflict and ambiguity. We explore the medical decision-makingprocess of physicians usingfunctional MRI. Twenty hospital physicians will be asked to make simulated medical decisions during fMRI acquisitions, with and without explicit budgetary constraints. We will compare the fMRI data between the 2 modalities.

ELIGIBILITY:
Inclusion Criteria:

* Hospital physicians
* working in the CHU of Montpellier

Exclusion Criteria:

* Contra indication to f-MRI

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital physicians
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Brain activation patterns measured by Functional magnetic resonance imaging | up to study completion, usually 2 weeks

SECONDARY OUTCOMES:
Level of role conflict, measured by the Kahn questionnaire (Kahn et al., 1964) | up tu study completion, usually 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire MERCIER, MD, PhD, Principal Investigator — University Montpellier Hospital

IPD SHARING:
Plan to Share IPD: No